CLINICAL TRIAL: NCT03955562
Title: Impact of Pedestrian Footbridges on Economic, Health and Educational Outcomes in Rural Communities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Yale University (Other); University of Notre Dame (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Evan Thomas, Associate Professor & Mortenson Endowed Chair in Global Engineering, and Director, Mortenson Center, University of Colorado, Boulder
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-0739
Record Dates: First submitted 2019-04-15; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Head of Household

STUDY DESIGN:
Intervention Model Description: The study will be a matched-cohort study, in which twelve bridge sites will be matched to twelve comparison sites. The bridge sites have been defined and identified by B2P staff in conjunction with government officials through a systematic needs assessment carried out in 2014. Of the twelve bridge sites that have been confirmed for the study, seven are located in the Southern Province, and five are located in the Western Province. Comparison sites were identified from a 2018 needs assessment carried out by B2P. As with the bridge sites, seven of the comparison sites are in the Southern Province and five are in the Western Province. The table of bridge and control sites with their respective districts and provinces can be found in Appendix A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Communities that receive a pedestrian footbridge.
  Interventions: Other: Footbridge
- Comparison (Experimental): Communities that do not receive a pedestrian footbridge.
  Interventions: Other: Comparison villages

INTERVENTIONS:
Other: Footbridge — Access to a pedestrian footbridge.
  Arms: Intervention
Other: Comparison villages — Villages that do not receive a footbridge.
  Arms: Comparison

SUMMARY:
Isolation caused by lack of transportation infrastructure affects almost every facet of life for the rural poor. Without adequate transportation access, families cannot access schools, health care, employment, or local markets to sell and buy goods. The World Bank estimates that nearly a billion people worldwide lack access to an all-season road within two kilometers, illustrating the scope of the problem, and the challenge of addressing it at scale.

Bridges to Prosperity (B2P) is a non-profit organization that builds footbridges to connect rural communities facing isolation to road networks and critical destinations and services. B2P has constructed more than 280 footbridges in 20 countries, an infrastructure intervention that is cost-effective, durable, and relatively simple to scale. B2P's field program in Rwanda started in 2012 and has led to the completion of 37 footbridges that have created new safe access for an estimated 225,000 people. Over the next five years, B2P plans to construct approximately 350 footbridges in Rwanda. This rapid program growth presents an unprecedented opportunity for rigorous investigation of the effects of new footbridges on a number of key economic, health, agricultural and education outcomes for rural communities.

As such, the research team has been brought on to carry out an impact evaluation of B2P-constructed footbridges in rural Rwanda. This protocol is for the first phase of the study and will focus on 12 footbridge sites and 12 comparison sites over the course of one year, while the larger study will encompass approximately 350 sites over the planned five-year construction period. The results of this first phase will inform the design of the larger study.

DETAILED DESCRIPTION:
The study will be a matched-cohort study, in which twelve bridge sites will be matched to twelve comparison sites. The bridge sites have been defined and identified by B2P staff in conjunction with government officials through a systematic needs assessment carried out in 2014. Of the twelve bridge sites that have been confirmed for the study, seven are located in the Southern Province, and five are located in the Western Province. Comparison sites were identified from a 2018 needs assessment carried out by B2P. As with the bridge sites, seven of the comparison sites are in the Southern Province and five are in the Western Province. The table of bridge and control sites with their respective districts and provinces can be found in Appendix A.

The minimum detectable effect analysis for outcomes of interest determined that, with these 24 sites, the investigators should survey representatives from 100 households in each treatment site (those receiving a bridge) and comparison site (those that will not). For both treatment sites and comparison sites, B2P will identify the impacted side - that which their assessment indicates would benefit the most from the bridge. Investigators will then obtain the administrative list of households from the umudugudu chief (village leader) or cell secretary for the village that is closest to the bridge on the impacted side. If the list consists of at least 100 households, investigators will randomly select the 100 households to visit from this list. If the village has fewer than 100 households, enumerators will visit all households in that village and then, from the list for the next closest village, randomly select the remaining number required to reach 100 households.

As part of the pilot study, investigators are testing an experimental method to determine which households to sample within a community. This method involves tracing satellite imagery of the relevant communities to derive a vector dataset of all the households in the area, from which investigators randomly select certain ones based upon an algorithm. This approach is intended to make the sampling more robust by reducing the opportunity to introduce human bias. The tracing of homesteads will be done using freely available Bing aerial imagery and the data generated will be contributed to OpenStreetMap (OSM), in accordance with the Bing imagery license for OpenStreetMap. While all the households traced will be uploaded to OSM and be publicly available, all subsequent analysis of which households are to be surveyed and survey results themselves will be kept in private on password-protected devices and will only be used for the purposes of the study.

The study will utilize a difference-in-difference empirical design. That is, it will compare changes over time in communities that receive a bridge against those that do not. This is recovered from a linear regression:

y_vt = a + β*Bridge_vt + E_vt In this equation, y_vt is some outcome of interest in community v at time t and Bridge_vt is an indicator of community v has a bridge at time t. Under the identification procedure described above, the coefficient β estimated in the above regression identifies the causal effect of bridge construction.

Based on the findings of Brooks and Donovan 2018, investigators are interested in exploring not only economic and agricultural outcomes but also using this larger opportunity to explore health and educational outcomes as well.

To utilize the difference-in-difference method, data is required for at least two points in time from all households in the study. Therefore, baseline surveys will be conducted before any bridges are built, followed by a second round of data from the same households after bridges are built, and a third round of data collection a year after the baseline. This will take place in both treatment communities and comparison communities.

The baseline survey will be conducted in February-March 2019. This corresponds with the main harvest period in Rwanda, allowing for the collection of specific information on agricultural outcomes while that information is still fresh in the minds of community members surveyed. The completion of bridges will begin in late February 2019 and continue through July 2019. A midline survey will be carried out in June-July 2019. And end-line data will be collected in February-March 2020. The same survey will be used at all three time points, thus allowing the testing of any differences that occur over time.

The survey will be carried out by trained enumerators fluent in Kinyarwanda on tablet computers. Once completed, the surveys will be uploaded directly to a secure server in the United States for analysis. A detailed list of the questions can be found in the attached survey.

As noted in the list of outcomes above, mid-upper arm circumference (MUAC) is one of the health outcomes of interest. MUAC is an easy body measurement that helps to monitor nutrition, and the nutritional status of children under five is a proxy indicator of the community's nutrition. However, MUAC is not used for children under six months of age because there are not established nutrition cutoff levels for this age group. With consent from the primary caregiver, MUAC will be measured for every child in the household who is between the ages of six months and five years. The instructions for this process are included in the survey.

In June 2019, cameras will be installed at the entrance to bridge crossings that will take pictures as individuals cross the bridges. This data will be analyzed to estimate bridge uses, allowing us to investigate the potential correlation between bridge use and economic, agricultural, health and educational benefits. The data from the cameras will be stored on local digital storage devices. The cameras will be locked in place. The camera data will be collected by study staff periodically and uploaded to secure, password protected databases. The pictures will be analyzed by computer and by study team review to count the number of users of the bridge. No personally identifiable information will be published in any form.

ELIGIBILITY:
Inclusion Criteria:

* Random selection of first 100 households in a village from administrative data
* Head of household in intervention and comparison villages

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Household food expenditure | 18 months
  Rwandan francs - percentage change from baseline Household representatives will be asked survey questions regarding the prices and quantities of consumption of food items to determine total household expenditure on food, including distinction between own-produced food and market purchases.
Household income | 18 months
  Rwandan francs - percentage change from baseline Household representatives will be asked survey questions regarding the income generating activities of adults in the household and the amount of income from each activity to determine total household income.
Household use of fertilizer | 18 months
  Yes/no - change in percentage Household representatives will be asked whether or not their household uses fertilizer when growing crops.
Monetary value of livestock | 18 months
  Rwandan francs - percentage change from baseline Household representatives will be asked survey questions regarding the types, quantities, and value of livestock their household owns.
Work outside of community | 18 months
  Yes/no - change in percentage yes/no) - change in percentage Household representatives will be asked survey questions regarding the location of work for adults in the household, and specifically whether individuals leave the community to work daily, seasonally or for longer periods of time.
Access to health care | 18 months
  Yes/no - change in percentage Household representatives will be asked whether or not household members have visited a health clinic in the last month.
Mid-upper arm circumference (MUAC) | 18 months
  Centimeters - percentage change from baseline With household representative's permission, the MUAC of children in the household between 6 months and 5 years will be measured using an MUAC tape.

SECONDARY OUTCOMES:
Child enrollment in school | 18 months
  Household representatives will be asked whether the children in the household are enrolled in school
Days of school missed | 18 months
  Household representatives will be asked how many days of school each child attending school missed in the past month
Access to prenatal care | 18 months
  If the household representative is pregnant or a household member under 18 is pregnant, the household representative will be asked if the pregnant woman or girl has visited a clinic for prenatal care during the current pregnancy.
Type of prenatal services received | 18 months
  If prenatal services have been received by a household member during a current pregnancy, the household representative will be asked what type of services were received.
Prenatal tetanus vaccination | 18 months
  If the household representative is pregnant or a household member under 18 is pregnant, the enumerator will request to see their vaccination card and document whether they have received their tetanus vaccine. If the card is not available or the respondent does not want to show the card, the enumerator will ask if the pregnant person has received their tetanus vaccine.
Child vaccination | 18 months
  For children under 5 years of age, the enumerator will ask to see their vaccination cards and, if available, document what vaccines the child has received. If not available or not made available, the enumerator will ask the household representative which vaccines the child has received.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Thomas, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Communities in Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No